CLINICAL TRIAL: NCT06646276
Title: A Randomized, Double Blind, Multicenter Phase 3 Trial of BMS-986489 (BMS-986012+Nivolumab Fixed Dose Combination) in Combination With Carboplatin Plus Etoposide vs Atezolizumab in Combination With Carboplatin Plus Etoposide as First-Line Therapy in Participants With Extensive-Stage Small Cell Lung Cancer (TIGOS).
Brief Title: A Study to Compare the Efficacy and Safety of BMS-986489 (BMS-986012+ Nivolumab Fixed Dose Combination) in Combination With Carboplatin Plus Etoposide to That of Atezolizumab With Carboplatin Plus Etoposide as First-Line Therapy in Participants With Extensive-Stage Small Cell Lung Cancer (TIGOS).
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA245-0001
Record Dates: First submitted 2024-10-16; First posted 2024-10-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Extensive-Stage Small Cell Lung Cancer
Keywords: BMS-986489; BMS-986012; Extensive-Stage Small Cell Lung Cancer; Etoposide; Carboplatin; Nivolumab; TIGOS; fucGM1; SCLC; ES-SCLC; atigotatug
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental)
  Interventions: Biological: BMS-986489 (BMS-986012+Nivolumab); Drug: Carboplatin; Drug: Etoposide
- Arm B (Active Comparator)
  Interventions: Biological: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Biological: BMS-986489 (BMS-986012+Nivolumab) — Specified dose on specified days
  Arms: Arm A
Biological: Atezolizumab — Specified dose on specified days
  Arms: Arm B
Drug: Carboplatin — Specified dose on specified days
Drug: Etoposide — Specified dose on specified days

SUMMARY:
The Purpose of the Study is to Compare the Efficacy and Safety of BMS-986489 (Anti-fucosyl-GM1+ Nivolumab Fixed Dose Combination) in Combination with Carboplatin plus Etoposide to that of Atezolizumab with Carboplatin plus Etoposide as First-Line Therapy in Participants with Extensive-Stage Small Cell Lung Cancer.

ELIGIBILITY:
Inclusion Criteria

* Participants must have diagnosis of Extensive-Stage Small Cell Lung Cancer (ES-SCLC).
* Participants must be Healthy enough to do their normal activities with little or no help based on the ECOG performance scale.
* Participants must have at least one tumor that can be measured using special imaging techniques like a CT scan or MRI at a site other than the brain and nervous system

Exclusion Criteria

* Participants have already received certain types of treatment for extensive stage small cell lung cancer
* Participants have certain health conditions, like spread of small cell lung cancer to the brain that are causing symptoms, certain lung diseases, heart diseases, infections, autoimmune diseases, other cancers, or a type of nerve damage called peripheral sensory neuropathy
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2025-02-25 (Actual); Primary Completion 2028-04-06 (Estimated); Study Completion 2031-09-05 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | Up to 5 years

SECONDARY OUTCOMES:
Time to definitive deterioration (TTDD)based on the LCSS ASBI defined as the time from randomization until a definitive clinically meaningful decline (≥ 10 point increase from baseline in LCSS ASBI score). | Up to 5 years
Number of participants with Adverse Events (AEs) | Up to 135 days after last treatment
Number of Participants with Serious Adverse Events (SAEs) | Up to 135 days after last treatment
Number of Participants with Adverse Events (AEs) leading to discontinuation and death | Up to 135 days after last treatment
Objective Response (OR) | Up to 5 years
Duration of Response (DOR) | Up to 5 years
Progression Free Survival (PFS) | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (184):
- United States (20):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Local Institution - 0283, Hot Springs, Arkansas
  - Florida Cancer Specialists - South, Fort Myers, Florida
  - Mid Florida Hematology and Oncology Center, Orange City, Florida
  - Florida Cancer Specialists - North, St. Petersburg, Florida
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital, Marietta, Georgia
  - Illinois Cancer Care, Peoria, Illinois
  - Local Institution - 0037, Minneapolis, Minnesota
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico
  - Duke Cancer Institute, Durham, North Carolina
  - Local Institution - 0232, Bismarck, North Dakota
  - Oncology Hematology Care, Cincinnati, Ohio
  - Sanford Cancer Center, Sioux Falls, South Dakota
  - SCRI Oncology Partners, Nashville, Tennessee
  - Texas Oncology - Central/South Texas, Austin, Texas
  - Local Institution - 0340, Dickinson, Texas
  - Texas Oncology - Northeast Texas, Tyler, Texas
  - Oncology & Hematology Associates of Southwest Virginia, Inc., Roanoke, Virginia
  - Swedish Cancer Institute - Edmonds, Edmonds, Washington
  - Swedish Medical Center, Seattle, Washington
- Argentina (5):
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Hospital Italiano de Buenos Aires, ABB, Buenos Aires F.D.
  - Local Institution - 0100, Buenos Aires, Buenos Aires F.D.
  - Clinica Adventista Belgrano, CABA, Buenos Aires F.D.
  - Instituto Médico Río Cuarto, Río Cuarto, Córdoba Province
- Australia (5):
  - GenesisCare - Campbelltown, Campbelltown, New South Wales
  - Nepean Hospital, Penrith, New South Wales
  - Gallipoli Medical Research Ltd, Brisbane, Queensland
  - Grampians Health, Ballarat Central, Victoria
  - St. John of God Murdoch Hospital, Murdoch, Western Australia
- Austria (4):
  - Medizinische Universität Graz, Graz, Styria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Kepler Universitätsklinikum, Linz
  - Landeskrankenhaus Rankweil, Rankweil
- Belgium (4):
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - UZ Gent, Ghent, Oost-Vlaanderen
  - VITAZ, Sint-Niklaas, Oost-Vlaanderen
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (7):
  - Hospital São Carlos, Fortaleza, Ceará
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul, Rio Grande do Sul
  - Clínica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - CIUSSS- saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - IUCPQ, Québec, Quebec
  - Centre intégré de santé et de services sociaux du Bas Saint-Laurent- Hôpital régional de Rimouski, Rimouski, Quebec
- Chile (5):
  - Oncocentro Apys, Viña del Mar, Región de Valparaíso
  - Orlandi Oncologia, Santiago, Santiago Metropolitan
  - Fundacion Arturo Lopez Perez (FALP), Santiago, Santiago Metropolitan
  - Pontificia Universidad Catolica de Chile, Santiago, Santiago Metropolitan
  - Bradfordhill, Santiago, Santiago Metropolitan
- China (23):
  - Peking University Cancer Hospital Beijing Cancer Hospital Beijing Institute for Cancer Research, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Wuhan Tongji Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province Tumor Hospital, Changchun, Jilin
  - Local Institution - 0235, Shenyang, Liaoning
  - Xi'an International Medical Center Hospital, Xi'an, Shaanxi
  - Shandong Cancer Hospital, Jinan, Shandong
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhongshan Hospital,Fudan University, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Linhai, Zhejiang
- Czechia (4):
  - Masarykuv onkologicky ustav, Brno, Brno-město
  - Nemocnice AGEL Ostrava - Vitkovice a.s., Ostrava, Ostrava Město
  - Fakultni Thomayerova nemocnice, Prague, Praha 4
  - Fakultni nemocnice Olomouc, Olomouc
- France (10):
  - Hôpital Arnaud de Villeneuve - CHU Montpellier, Montpellier, Hérault
  - Chu Grenoble Alpes, La Tronche, Isère
  - CHU Lille - Institut Coeur Poumon, Lille, Nord
  - L Hopital Nord Ouest, Gleizé, Rhône
  - Centre Hospitalier Lyon Sud, Pierre-Bénite, Rhône
  - Centre Hospitalier Intercommunal de Créteil, Créteil, Val-de-Marne
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Institut Curie, Paris
  - Centre Hospitalier de Cornouaille Quimper - Concarneau, Quimper
- Germany (9):
  - Krankenhaus Nordwest GmbH, Frankfurt am Main, Hesse
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Klinikum Köln-Merheim, Cologne, North Rhine-Westphalia
  - Krankenhaus Martha-Maria Halle-Dölau, Halle, Saxony-Anhalt
  - Zentralklinik Bad Berka, Bad Berka, Thuringia
  - Asklepios Klinik Gauting GmbH, Gauting
  - LungenClinic Grosshansdorf, Großhansdorf
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg
  - Robert Bosch Krankenhaus GmbH, Stuttgart
- Greece (5):
  - Errikos Dunant Hospital Center, Athens, Attikí
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attikí
  - "Theagenio" Cancer Hospital of Thessaloniki, Thessaloniki, Kentrikí Makedonía
  - European Interbalkan Medical Center, Thessaloniki, Thessaloníki
  - University General Hospital of Larissa, Larissa, Thessalía
- India (5):
  - Manipal Hospitals, Bengaluru, Karnataka
  - Local Institution - 0278, New Delhi, National Capital Territory of Delhi
  - Meenakshi Mission Hospital and Research Centre, Madurai, Tamil Nadu
  - Mahamana Pandit Madan Mohan Malviya Cancer Centre, Varanasi, Uttar Pradesh
  - Netaji Subhas Chandra Bose Cancer Hospital, Kolkata, West Bengal
- Italy (7):
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale, Napoli, Campania
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Lombardy
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - AO Santa Maria della Misericordia, Perugia, Umbria
  - Casa di Cura Dott. Pederzoli, Peschiera del Garda, Verona
  - IRCCS Azienda Ospedaliero-Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna
  - Istituto Europeo di Oncologia IRCCS, Milan
- Japan (18):
  - National Hospital Organization Shikoku Cancer Center, Matsuyama, Ehime
  - Kurume University Hospital, Kurume, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cardiovascular and Respiratory Center, Yokohama, Kanagawa
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Nara Medical University Hospital, Kashihara, Nara
  - Kurashiki Central Hospital, Kurashiki, Okayama-ken
  - Kansai Medical University Hospital, Hirakata, Osaka
  - Kindai University Hospital- Osakasayama Campus, Ōsaka-sayama, Osaka
  - Osaka Medical and Pharmaceutical University Hospital, Takatsuki, Osaka
  - Saitama Medical University International Medical Center, Hidaka, Saitama
  - Saitama Prefectural Cancer Center, Ina-machi, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Koto, Tokyo
  - Fukushima Medical University, Fukushima
- Malaysia (3):
  - Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Sarawak General Hospital, Kuching, Sarawak
- Mexico (3):
  - Local Institution - 0146, Guadalajara, Jalisco
  - Local Institution - 0147, Monterrey, Nuevo León
  - Unidad Médica Onco-hematológica, Puebla City
- Netherlands (3):
  - Amsterdam UMC, locatie VUmc, Amsterdam, North Holland
  - Ziekenhuis Rijnstate, Arnhem
  - University Medical Center Groningen, Groningen
- Poland (5):
  - Przychodnia Lekarska KOMED, Konin, Greater Poland Voivodeship
  - Centrum Medyczne Pratia Poznań, Poznan, Greater Poland Voivodeship
  - Szpital Specjalistyczny w Prabutach Spolka z o.o., Prabuty, Pomeranian Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Łódź Voivodeship
- Romania (7):
  - SC Memorial Healthcare International SRL, Bucharest, București
  - Institutul Oncologic Bucuresti "Prof. Dr. Alexandru Trestioreanu", Bucharest, București
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Institutul Oncologic Cluj, Cluj-Napoca
  - S.C. Centrul de Oncologie Euroclinic S.R.L., Iași
  - Institutul Regional de Oncologie, Iași
- South Korea (6):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Seoul National University Bundang Hospital, Seongnam, Kyǒnggi-do
  - Ajou University Hospital, Suwon, Kyǒnggi-do
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Asan Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Keimyung University Dongsan Hospital, Daegu, Taegu-Kwangyǒkshi
- Spain (10):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [Cataluña]
  - Hospital de la Santa Creu i Sant Pau, Barcelona, Catalunya [Cataluña]
  - Hospital Universitario de Jaen, Jaén, Jaén
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Switzerland (3):
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Winterthur, Winterthur
  - UniversitätsSpital Zürich, Zurich
- Turkey (Türkiye) (5):
  - T.C. Saglik Bakanligi - Izmir Il Saglik Mudurlugu Cigli Bolge Egitim Hastanesi, Çiğli, İzmir
  - Local Institution - 0154, Adana
  - Gulhane Egitim Arastirma Hastanesi, Ankara
  - Atatürk Göğüs Hastalıkları Ve Göğüs Cerrahisi Eğitim Araştırma Hastanesi, Ankara
  - Istanbul Medeniyet University, Istanbul
- United Kingdom (4):
  - James Cook University Hospital, Central Middlesbrough, Middlesbrough
  - Aberdeen Royal Infirmary, Aberdeen
  - The Christie NHS Foundation Trust, Manchester
  - The Clatterbridge Cancer Centre, Metropolitan Borough of Wirral

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol-Myers Squibb's data sharing policy and process can be found at: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06646276.html